CLINICAL TRIAL: NCT05783505
Title: PRevention of pAtient's agItation and Enhancement of Their SafEty (PRAISE): Improving Intensive Care Treatment Using a Multicomponent Pharmacological Intervention
Brief Title: A Multicomponent Intervention Program to Prevent and Reduce ICU Agitation and Physical Restraint Use
Acronym: PRAISE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-16133
Record Dates: First submitted 2023-01-08; First posted 2023-03-24 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Agitation,Psychomotor
Keywords: ICU; Agitation; Physical Restraints; Non-pharmacologic interventions; Dexmedetomidine
MeSH Terms: conditions — Psychomotor Agitation

STUDY DESIGN:
Intervention Model Description: Multicenter stepped wedge cluster randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Experimental): Multicomponent intervention program
  Interventions: Other: Multicomponent intervention program
- Control group (No Intervention): Standard care

INTERVENTIONS:
Other: Multicomponent intervention program — Non-pharmacological interventions combined with goal directed sedation using dexmedetomidine if needed
  Arms: Treatment group

SUMMARY:
Despite deleterious effects, physical restraints are still commonly used in (expected to become) agitated patients in Dutch ICUs (20-25%). This study aims to determine the effectiveness of a person-centered multicomponent intervention (MCI) program consisting of non-pharmacological interventions combined with goal directed light sedation using dexmedetomidine compared to the old standard of care including physical restraints in (expected to become) agitated adult ICU patients.

DETAILED DESCRIPTION:
Applying physical restraints (PR) has detrimental short- and long-term effects on patients and is increasingly seen as inhumane and outdated. Nonetheless, PR are still used in approximately 20-25% of all patients during their intensive care unit (ICU) stay in the Netherlands. The aim of this study is to determine the effectiveness of a person-centered multicomponent intervention (MCI) program consisting of non-pharmacological interventions combined with goal directed light sedation using dexmedetomidine compared to the old standard of care including physical restraints on short- and long-term outcomes and healthcare costs in (expected to become) agitated adult ICU patients.

ELIGIBILITY:
Inclusion criteria:

* Adult ICU patients (aged ≥18) with an expected ICU stay of >24 hours
* Patients who are (expected to become) agitated within the first 14 days of their ICU admission

Exclusion criteria:

* Contra indication for dexmedetomidine use (i.e., AV-block grade 2 or 3 unless a pacemaker is present, uncontrolled hypotension, acute cerebrovascular condition or known/suspected hypersensitivity);
* Neurological patients with an (expected risk of) increased intracranial pressure;
* An intoxication as a result of drug abuse (e.g., ethanol, γ-Hydroxybutyrate, opioids, benzodiazepines);
* Support with Extracorporeal Membrane Oxygenation (ECMO);
* Difficult airway (e.g., a Cormack and Lehane laryngoscopy grade 4 view or a tumor causing airway obstruction);
* A high risk of physical aggression towards healthcare professionals;
* No consent for long term follow up in the MONITOR-IC study;
* Not able to read or understand the Dutch language and no relatives able to assist;
* Enrolment in other sedation studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
ICU-free days | 28 days

SECONDARY OUTCOMES:
Incidence rate of accidentally removed medical devices | 14 days
Incidence rate of (self-extubation induced) reintubations | 14 days
Days with delirium | 14 days
  Assessed using the Intensive Care Delirium Screening Checklist (ICDSC), Confusion Assessment Method for the ICU (CAM-ICU), or the Delirium Observation Screening scale for the ward (DOS)
Days with coma | 14 days
  Assessed using the Richmond Agitation and Sedation Scale (RASS)
Number of delirium- and coma-free days | 14 days
Days with physical restraints | 14 days
Days with dexmedetomidine (and total administered dose) | 14 days
Dexmedetomidine related adverse events (e.g., hypotension, bradycardia) that required intervention | 14 days
Days with propofol (and total administered dose) | 14 days
Duration of mechanical ventilation in days | up to 180 days
Hospital length of stay in days | up to 180 days
Mortality | at 28 days, 3 months and 12 months
Physical outcome | at ICU admission, 3, 12 and 24 months
  E.g., fatigue, frailty, new or worsened physical problems, assessed using validated questionnaires
Mental outcome | at ICU admission 3, 12 and 24 months
  E.g., post traumatic stress disorder (PTSD), anxiety, depression, assessed using validated questionnaires
Cognitive outcome | at 3, 12 and 24 months
  E.g., cognitive impairment, assessed using a validated questionnaire
Quality of life | at ICU admission, 3, 12 and 24 months
  Assessed using a validated QoL questionnaire
Cost-effectiveness | 12 months
  Measured by cost per Quality-Adjusted Life Year (QALY)

OTHER OUTCOMES:
Incidence rate of falls out of bed | 14 days
A secondary Bayesian analysis of the trial including heterogeneity of treatment effect | To be conducted within one year after study completion
  A secondary Bayesian analysis of the trial including heterogeneity of treatment effect

CONTACTS AND LOCATIONS:
Overall Officials: Bram Tilburgs, PhD, Principal Investigator — Radboud University Medical Center; Mark van den Boogaard, PhD, Study Director — Radboud University Medical Center
Locations (5):
- Netherlands (5):
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Bravis Ziekenhuis, Bergen op Zoom
  - Amphia Ziekenhuis, Breda
  - Elkerliek Ziekenhuis, Helmond
  - VieCuri Medisch Centrum, Venlo

IPD SHARING:
Plan to Share IPD: Yes
upon reasonable request

REFERENCES:
- [Derived] Kooken RWJ, Tilburgs B, Ter Heine R, Ramakers B, van den Boogaard M; PRAISE study group. A multicomponent intervention program to Prevent and Reduce AgItation and phySical rEstraint use in the ICU (PRAISE): study protocol for a multicenter, stepped-wedge, cluster randomized controlled trial. Trials. 2023 Dec 11;24(1):800. doi: 10.1186/s13063-023-07807-x. PMID 38082351